CLINICAL TRIAL: NCT06108895
Title: Ilioinguinal Iliohypogastric Nerve Block Compared to Intrathecal Morphine as Adjunct to Spinal Anesthesia for Cesarean Section: Randomized Controlled Trail
Brief Title: Ilioinguinal Iliohypogastric Nerve Block as Adjunct to Spinal Anesthesia for Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Sobhy Mohamed Basyouni, professor of anethesia and critical care, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 36264PR333/9/23
Record Dates: First submitted 2023-10-20; First posted 2023-10-31 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Cesarean Section; Post Operative Pain
Keywords: Ilioinguinal/Iliohypogatric; Peripheral Nerve Block; Cesarean Section
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Ninty parturients who had normal singleton pregnancy scheduled for elective lower segment cesarean section through a Pfannensteil incision under spinal anesthesia will be recruited in the study. They will be randomly divided into three equal groups; Group C, control group who will receive spinal anesthesia; Group M who will receive spinal anesthesia with intrathecal morphine, and group I who will receive spinal anesthesia and IINB
Who Masked: Outcomes Assessor
Masking Description: A single researcher who will be blinded to groups will be responsible for all measurements and data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C, control group (No Intervention): it will receive intrathecal 12.5 mg (2.5ml) hyperbaric bupivacaine 0.5%.
- Group I (Active Comparator): it will receive intrathecal 12.5 mg (2.5ml) hyperbaric bupivacaine 0.5% plus bilateral ultrasound guided IINB after surgery.
  Interventions: Other: ilio-inguinal/ilio-hypogastric nerve block (IINB)
- Group M (Active Comparator): it will receive intrathecal 12.5 mg hyperbaric bupivacaine 0.5% plus 200 mcg morphine in 2.5ml solution.
  Interventions: Other: intrathecal morphine

INTERVENTIONS:
Other: ilio-inguinal/ilio-hypogastric nerve block (IINB) — Ultrasound-guided IINBs will be performed by scanning the anterior abdominal wall superior and medial to the anterior superior iliac spine in a line between the anterior superior iliac spine and umbilicus using a linear probe (4-12hertz). Ilioinguinal and iliohypogastric nerves will be identified in the plane between internal oblique muscle and transversus abdominis muscle. After negative aspiration of blood, 20 ml plain bupivacaine 0.25% plus 4mg dexamesathone will be injected. The same technique will be performed in the other side.
  Arms: Group I
Other: intrathecal morphine — 200 mcg morphine intrathecally with bupivacaine
  Arms: Group M

SUMMARY:
The aim of the present controlled randomized study is to compare between ilioinguinal/iliohypogastric nerve block (IINB) and morphine as adjuncts to spinal anesthesia for cesarean section regarding quality of post-operative analgesia. The researchers will compare between the following groups: Group C, control group; will receive intrathecal 12.5 mg hyperbaric bupivacaine 0.5%, Group I; will receive intrathecal 12.5 mg hyperbaric bupivacaine 0.5% plus bilateral ultrasound guided IINB, and Group M; will receive intrathecal 12.5 mg hyperbaric bupivacaine 0.5% plus 200 mcg morphine to answer the question: Could IINB be an alternative to intrathecal morphine during spinal anesthesia for cesarean section ?.

DETAILED DESCRIPTION:
Ninty full term healthy non laboring parturient between 21 and 40 years of age who had normal singleton pregnancy scheduled for elective lower segment cesarean section through a Pfannensteil incision under spinal anesthesia will be recruited in the study after obtaining an informed written consent.

During the preoperative visit, parturient will be explained how to use pain numeric rating scale (PNRS), post-operative nausea and vomiting (PONV) intensity scale, and Likert 4 point satisfaction scale.

The participated parturients will be divided randomly using a computer generated random table into three equal groups thirty patient each; C, I, and M. Group C, control group; will receive intrathecal 12.5 mg hyperbaric bupivacaine 0.5% (2.5ml). Group I; will receive intrathecal 12.5 mg hyperbaric bupivacaine 0.5% (2.5ml) plus bilateral ultrasound guided IINB at the end of surgery after suturing and dressing the wound. Group M; will receive intrathecal 12.5 mg hyperbaric bupivacaine 0.5% plus 200 mcg morphine in 2.5ml solution.

In the morning of surgery; all participants will be administered IV infusion of 40mg pantoprazole diluted in 500 ml of lactated ringer over 30 min. Pulse oximeter, ECG and noninvasive blood pressure will be connected to the participant on arrival to the operating room. Spinal anesthesia will be given in the sitting position under complete aseptic precaution at L3-4 or L4-5 subarachnoid space with a 25 or 27 gauge Sprotte spinal needle. Loss of Light touch sensation on the mid-clavicular line below T 7 will be considered adequate for start of surgery.

Ultrasound guided IINB will be performed by scanning the anterior abdominal wall superior and medial to the anterior superior iliac spine in a line between the anterior superior iliac spine and the umbilicus using a linear probe (4-12hertz). Ilioinguinal and iliohypogastric nerves will be identified in the plane between the internal oblique muscle and the transversus abdominis muscle. After negative aspiration of blood; 20 ml plain bupivacaine 0.25% plus 4mg dexamesathone will be injected. The same technique will be performed on the other side.

All parturients will be given IV acetaminophen 1g/8h and IV Lornoxicam 8mg/12h. Rescue IV 3mg morphine will be given if pain score ≥ 4 is reported during the first post-operative 24 hours.

The following parameters will be recorded; demographics, vital signs, and quality of postoperative analgesia using the PNRS, ranging from 0 (no pain) to 10 (severe pain); at rest and during movement in the following time points: Time 0; end of surgery (T0), T1 (4 hours after surgery), T2 (6 hours after surgery), T3 (12 hours after surgery), T4 (18 hours after surgery), T 5 (24 hours after surgery), T 6 (36 hours after surgery), T 7 (48 hours after surgery), and T8 (72 hours after surgery), total amount of rescue morphine during the first 24h after surgery, time to first ambulation, and complications including pruritus, PONV using the PONV intensity score, sedation using Ramsey sedation score, respiratory depression (respiratory rate ≤ 8/min), and complications related to IINB as improper block, pain, hematoma or infection at the site of injection. Patient's satisfaction will be assessed 72 hours after surgery using Likert 4 point scale. A single researcher who will be blinded to groups will be responsible for all measurements and data collection.

ELIGIBILITY:
Inclusion Criteria:

* Ninty full term healthy non laboring parturient between 21 and 40 years of age who had normal singleton pregnancy scheduled for elective lower segment cesarean section through a Pfannensteil incision under spinal anesthesia will be recruited in the study after obtaining an informed written consent

Exclusion Criteria:

* if they were using any medications other than prenatal vitamins, requiring an emergent cesarean section, having antepartum bleeding, diabetes mellitus, preeclampsia, eclampsia, history of substance abuse, or progressive neurological disease, having contraindication to spinal anesthesia as allergy to the study medications or infection at the site of injection, or they refused to participate in the study.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — full term healthy non laboring parturient between 21 and 40 years of age who had normal singleton pregnancy scheduled for elective lower segment cesarean section through a Pfannensteil incision under spinal anesthesia will be recruited in the study after obtaining an informed written consent
Enrollment: 90 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
pain numeric rating score at rest | Time 0: at end of surgery (T0); then 4hours (T1), 6hours (T2), 12hours (T3), 18hours (T4), 24hours (T5), 36hours (T6), 48hours (T7), and 72hours (T8) after surgery
  Patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. 0 represents 'no pain at all' where as 10 represents 'the worst pain ever possible'.
pain numeric rating score during movement | Time 0: at end of surgery (T0); then 4hours (T1), 6hours (T2), 12hours (T3), 18hours (T4), 24hours (T5), 36hours (T6), 48hours (T7), and 72hours (T8) after surgery
  Patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. 0 represents 'no pain at all' where as 10 represents 'the worst pain ever possible'.
total amounts of rescue morphine | at the end of the first 24 hours after surgery
  total amount of intravenous rescue morphine
time to first ambulation | the time the patient left the bed
  number of hours from end of surgery to the time the pateint left the bed
complications | during the first 72 hours after surgery
  pruritus, post-operative nausea and vomiting (PONV) using the PONV intensity score, sedation using Ramsey sedation score, respiratory depression (respiratory rate ≤ 8/min.), and complication related to IINB as improper block, pain, hematoma or infection at the site of injection.

SECONDARY OUTCOMES:
Patients' satisfaction | 72 hours after surgery
  Likert 4 point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Basyouni, MD, Principal Investigator — Anesthesia, intensive care, and pain management department; Tanta University, Egypt
Locations (1):
- Tanta University, Tanta, Gharbiah, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD will be shared as an excel sheet is requested by the other researcher

REFERENCES:
- [Background] DeSousa KA, Chandran R. intrathecal morphine for postoperative analgesia: current trends. World J Anesthesiol 2014; 3(3): 191-202
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] Hu P, Harmon D, Frizelle H. Ultrasound guidance for ilioinguinal/iliohypogastric nerve block: a pilot study. Ir J Med Sci. 2007 Jul-Sep;176(2):111-5. doi: 10.1007/s11845-007-0017-y. Epub 2007 Mar 20. PMID 17570011
- [Background] Krishnegowda S, Pujari VS, Doddagavanahalli SRC, Bevinaguddaiah y, Parate LH.A Randomized Control Trial on the Efficacy of Bilateral Ilioinguinal Iliohypogastric Nerve Block and Local Infiltration for Post Caesarean Delivery Analgesia. Journal of Obstetric Anaesthesia and Critical Care 2020; 10(1): 32-37
- [Result] Aasbo V, Thuen A, Raeder J. Improved long-lasting postoperative analgesia, recovery function and patient satisfaction after inguinal hernia repair with inguinal field block compared with general anesthesia. Acta Anaesthesiol Scand. 2002 Jul;46(6):674-8. doi: 10.1034/j.1399-6576.2002.460607.x. PMID 12059890
- [Result] Elahwal L, Elrahwan S, Elbadry AA. Ilioinguinal and Iliohypogastric Nerve Block for Acute and Chronic Pain Relief After Caesarean Section: A Randomized Controlled Trial. Anesth Pain Med. 2022 Mar 27;12(2):e121837. doi: 10.5812/aapm.121837. eCollection 2022 Apr. PMID 35991778